CLINICAL TRIAL: NCT01886183
Title: Effects of Training in a Virtual Environment on the Motor Function,Postural Control and Quality of Life in Chronic Stroke Patients: A Randomized Controlled Trial
Brief Title: Effects of Training in a Virtual Environment in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPNEC005
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: Postural Balance; Virtual Reality Exposure Therapy; Gait; Stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality Training (Experimental): The virtual reality training will be done by experimental group with ten games of Nintendo Wii Fit.
  Interventions: Other: Virtual Reality Training
- Control group: Physical Therapy (Active Comparator): The Control Group will be trained by conventional Physical Therapy exercises.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Virtual Reality Training — The participants of the study will be trained 8 balance games during 14 sessions
  Arms: Virtual Reality Training
Other: Physical Therapy — Patients of the control group will be trained with balance exercises.
  Other Names: Control group
  Arms: Control group: Physical Therapy

SUMMARY:
The objective of this work will be compare the effects of two balance training programs, one Nintendo Wii Fit-based and the other traditionally-based without the use of a gaming system, on the (1) motor function, (2) cognition, (3) balance and (4) gait in chronic stroke patients. It is a prospective, single blinded, randomized clinical trial performed at Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. Forty patients will be randomly assigned in control and experimental group, 20 each one.

DETAILED DESCRIPTION:
The objective of this work is to compare the effects of two balance training programs, one Nintendo Wii Fit-based and the other traditionally-based without the use of a gaming system, motor function, balance and quality of life in chronic stroke patients. It is a prospective, single-blinded, randomized clinical trial performed at Center of Research of the courses of Speech Therapy, Physical Therapy and Occupational Therapy of São Paulo University. Forty chronic stroke patients are randomly in control and experimental group, 20 each one. Both groups conduct 14 training sessions, twice a week, for seven weeks. Each session will consist a 30 minute-global-exercise series including stretching, muscle strength and axial mobility exercises. After this, both groups will performed more 30 minutes of balance training: the control group will performed balance exercises without external cues, visual or auditory feedbacks or cognitive stimulations; the experimental group will performed the balance training with 8 Wii Fit games which stimulate motor and cognitive functions. The main outcome measures will be: (1) the lower limb subscale of the Fugl-Meyer Assessment (FMA-LE); (2); Balance Evaluation Systems Test (BESTest);(3) the Stroke-Specific Quality of Life (SS-QOL); (4) 6- minute walk test (6MWT) and (5) The limits of stability (LOS).

ELIGIBILITY:
Inclusion Criteria:

* hemiparetic status resulting from a single stroke at least 6 months earlier;
* the ability to walk 10 m independently with or without an assistive device;
* the absence of a musculoskeletal condition that could potentially affect the ability to walk safely;
* the absence of serious visual impairment or a hearing disorder;
* power of at least grade 3 in the hemiplegic lower extremity;
* able to understand and follow simple instructions.

Exclusion Criteria:

* a Montreal Cognitive Assessment (MoCA) score of < 20;
* severe dementia or aphasia;
* hemispatial neglect, ataxia or any other cerebellar symptom;
* inability to stand without minimal assist;
* Impaired vision
* Uncontrollable medical complications
* participation in other studies or rehabilitation programs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The lower limb subscale of the Fugl-Meyer Assessment (FMA-LE) | up to 2 months
  FMA-LE is a subscale measuring lower limb motor recovery. It examines movement and coordination of the hip, knee, and ankle in the supine, sitting, and standing positions. Each item is scored on a 3-point scale (0, cannot perform; 1, partially performs; 2, performs fully). The score range is 0 to 34, with higher scores indicating better lower limb motor performance

SECONDARY OUTCOMES:
Balance Evaluation Systems Test (BESTest) | Up 2 months
  Balance Evaluation Systems Test (BESTest) measures balance. It includes 36 items that evaluate performance of 6 balance systems: biomechanical constraints, stability limits/verticality, anticipatory postural adjustments, postural responses, sensory orientation, and stability in gait.
6-minute walk test | Up to 2 months
  The 6MWT is a practical simple test. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). The 6MWT has been used as a measure of functional status of patients.
Stroke speciﬁc quality of life scale | Up to 2 months
  Stroke Speciﬁc Quality of Life Scale is a self-report assessment that includes 12 stroke speciﬁc subscales with 49 items. The Stroke Speciﬁc Quality of Life Scale attempts to capture the domains of stroke speciﬁc QOL that are insufficiently assessed with generic QOL measures. The 12 subscales, which are unidimensional, are Energy, Family Role, Language, Mobility, Mood, Personality, Self-Care, Social Roles, Thinking, Upper Extremity Function, Vision, and Work-Productivity. Participants responded to each item on a 5-point scale. Domain scores are the averages of the item scores, and the total score is the average of the domain scores. All summary scores therefore range from 1 to 5. Higher scores indicate better function.
Limits of Stability | Up to 2 months
  The Limits of Stability subtest quantifies the maximum distance a person can intentionally displace their center of pressure (COP) from start position of midline COP centered over the base of support to eight targets. Location and movement of the COP was indicated by a cursor display projected on a screen in front of the subject. As targets were highlighted, the subject was to move the COP cursor quickly and accurately as possible towards a target located on the Limits of Stability perimeter and hold position as close to the target as possible. The parameters include COP movement velocity and directional control (% to target).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PT, PhD, Study Director — University of Sao Paulo; Tatiana P Oliveira, PhD student, Principal Investigator — University of Sao Paulo; Camila S Miranda, Ms Student, Principal Investigator — University of Sao Paulo
Locations (1):
- Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo, São Paulo, Brazil